CLINICAL TRIAL: NCT03242226
Title: The Effect of +3.00ADD on Myopia Progression in Chinese Children: A Cluster Randomized Controlled Clinical Trial
Brief Title: The Effect of +3.00ADD on Myopia Progression in Chinese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-OPH-001
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Myopia
Keywords: +3.00ADD; single vision spectacle
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two spectacles (Experimental)
  Interventions: Device: two spectacles
- single vision spectacles (Active Comparator)
  Interventions: Device: single vision spectacles

INTERVENTIONS:
Device: two spectacles — single-vision spectacles for distant vision, and +3.00ADD spectacle for near vision
  Arms: two spectacles
Device: single vision spectacles — Wear single vision spectacle only
  Arms: single vision spectacles

SUMMARY:
The purpose of this study is to evaluate the effect of +3.00ADD vs single vision spectacle on the progression of myopia in children. Many studies applying bifocals or multifocal spectacles to intervene the progression have been carried out based on the idea that myopia was caused by excessive accommodation, however, the effect was limited. The possible reason is that bifocal or multifocal spectacles still not fully adjust the accommodative error in myopia children.

DETAILED DESCRIPTION:
The optical intervention has been extensively explored for the intervention of myopia progression.

Based on the theory that myopia was caused by the excessive accommodative, bifocal or multifocal spectacles for slowing the progression of myopia have been fully studied. Although some studies' results showed statistically significant for slowing myopia progression with multifocal spectacles, few had clinically meaningful, even in children with high accommodative lag or near-point esophoria. The investigators think that the possible reason for this clinical un-meaningful maybe that daily wearing bifocal or multifocal spectacles still not fully adjust the accommodative error in children.

The aim of this randomized clinical trial is to evaluate myopic progression in children using two spectacles (single-vision spectacles for distant vision, and +3.00ADD spectacle for near vision), compared with control subjects wearing one spectacles (single-vision spectacles). Myopia progression quantified by changes in axial length (AL) and cycloplegic spherical equivalent refraction will be monitored for 3 years. The spectacles for intervention group children will be adjusted based on the cycloplegic spherical equivalent and the extent of accommodation lag for schedule time.

ELIGIBILITY:
Inclusion criteria

1. Children who are aged 8 to 12 years (grade 3 and grade 4) from Huadu district of Guangzhou in China.
2. Refractive error meeting all the following, obtained by cycloplegic autorefraction: spherical equivalent -1.00 to -6.00D in both eyes, astigmatism ≤2.00 D in both eyes, and spherical equivalent anisometropia ≤1.50 D.
3. The best corrected visual acuity is ≥ 6/9.5
4. The parents are willing to provide consent to participation in the study, and the children are willing to wear the only provided spectacles

Exclusion criteria

1. Children who are allergy to tropicamide or topical anesthetic drugs.
2. Children who had other eye diseases that cause the visual impairment including strabismus, amblyopia, ocular surface related disease, cataract, traumas, ocular fundus diseases, and ocular surgery.
3. Children who were wearing rigid gas permeable contact lenses, progressive-addition lenses, bifocal spectacles lens, Peripheral defocus modifying contact lenses;
4. Children who are receiving visual function training.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent refraction (SER) change | 3 years
  SE was measured by autorefractometer with cycloplegic once a year at scheduled time

SECONDARY OUTCOMES:
axial length | 3 years
  Axial length is measured by IOMaster once a year at scheduled time
corneal curvature | 3 years
  Corneal curvature is measured by IOMaster once a year at scheduled time
binocular vision | 3 years
  the binocular vision was measured by an ophthalmologist every six month at scheduled time.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi LIU, MD,PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yangfa ZENG, MD,Master, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yet-san University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided